CLINICAL TRIAL: NCT06679075
Title: Clinical and Radiographic Evaluation of Propolis As a Hemostatic Agent for Pulpotomy of Mature Permanent Molars with Irreversible Pulpitis Using Two Different Dressing Materials; a Randomized Clinical Trial
Brief Title: Clinical and Radiographic Evaluation of Propolis As a Hemostatic Agent for Pulpotomy of Mature Permanent Molars with Irreversible Pulpitis Using Two Different Dressing Materials
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Misr International University (Other)
Responsible Party: Principal Investigator, Omar Hisham Selim, Master's of Endodontics Candidate, Misr International University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MIU-IRB-2324-047
Record Dates: First submitted 2024-11-06; First posted 2024-11-07 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Irreversible Pulpitis; Pulpitis; Pulpitis - Irreversible
Keywords: Pulpotomy; Vital Pulp Therapy; Adult Pulpotomy; Irreversible Pulpitis; Hemostasis; Hemostatic Agent; Propolis; MTA; Bioceramic; Full Pulpotomy; Mineral Trioxide Aggregate; Moderate Pulpitis; Severe Pulpitis; Mature Permanent Molars
MeSH Terms: conditions — Pulpitis | interventions — Pemetrexed

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Propolis + Bioceramic putty (Experimental): Adult permanent molars diagnosed with irreversible pulpitis to be treated with full pulpotomy using propolis as a hemostatic agent and bioceramic putty as a dressing material.
  Interventions: Procedure: Full pulpotomy using propolis and bioceramic putty
- Propolis + MTA (Experimental): Adult permanent molars diagnosed with irreversible pulpitis to be treated with full pulpotomy using propolis as a hemostatic agent and MTA as a dressing material.
  Interventions: Procedure: Full pulpotomy using Propolis and MTA
- Sodium hypochlorite + bioceramic putty (Experimental): Adult permanent molars diagnosed with irreversible pulpitis to be treated with full pulpotomy using sodium hypochlorite (NaOCl) as a hemostatic agent and bioceramic putty as a dressing material.
  Interventions: Procedure: Full pulpotomy using sodium hypochlorite and bioceramic putty
- Sodium hypochlorite + MTA (Active Comparator): Adult permanent molars diagnosed with irreversible pulpitis to be treated with full pulpotomy using sodium hypochlorite (NaOCl) as a hemostatic agent and MTA as a dressing material
  Interventions: Procedure: Full pulpotomy using sodium hypochlorite and MTA

INTERVENTIONS:
Procedure: Full pulpotomy using propolis and bioceramic putty — Full Pulpotomy for participants with mature adult molars diagnosed with irreversible pulpitis; using Propolis as a hemostatic agent and bioceramic putty as a dressing material
  Arms: Propolis + Bioceramic putty
Procedure: Full pulpotomy using Propolis and MTA — Full Pulpotomy for participants with mature adult molars diagnosed with irreversible pulpitis; using Propolis as a hemostatic agent and MTA as a dressing material
  Arms: Propolis + MTA
Procedure: Full pulpotomy using sodium hypochlorite and bioceramic putty — Full Pulpotomy for participants with mature adult molars diagnosed with irreversible pulpitis; using sodium hypochlorite (NaOCl) as a hemostatic agent and bioceramic putty as a dressing material
  Arms: Sodium hypochlorite + bioceramic putty
Procedure: Full pulpotomy using sodium hypochlorite and MTA — Full Pulpotomy for participants with mature adult molars diagnosed with irreversible pulpitis; using sodium hypochlorite (NaOCl) as a hemostatic agent and MTA as a dressing material.
  Arms: Sodium hypochlorite + MTA

SUMMARY:
The goal of this clinical trial is to assess the effectiveness of propolis as a hemostatic agent in pulpotomy for adult permanent molars, compared to sodium hypochlorite (NaOCl). It also examines how bioceramic putty performs against mineral trioxide aggregate (MTA) in vital pulp therapy for cases of irreversible pulpitis.

Participants will be divided into four groups (15 patients each):

* Propolis + bioceramic putty
* Propolis + MTA
* Sodium hypochlorite + bioceramic putty
* Sodium hypochlorite + MTA The Investigator will record the bleeding time and postoperative pain will be recorded. The researcher will assess the clinical and radiographic outcomes for success at 1, 3, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Participants of both genders falling within the age range of 20 to 45 years.
* Presence of vital mature permanent molars diagnosed as mild or severe irreversible pulpitis per Wolter's classification.
* Confirmation of vital bleeding pulp tissue in all canals following complete pulpotomy.

Exclusion Criteria:

* Non-vital teeth.
* Teeth with Immature roots.
* Uncontrolled pulpal bleeding persisting beyond 10 minutes post-application of sodium hypochlorite as a hemostatic agent.
* Insufficient bleeding post-pulp exposure, indicative of pulp degeneration.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Clinical and radiographic success rate | 1, 3, 6 months
  Success rate of full pulpotomy procedure using different hemostatic agents and different dressing materials using the clinical and radiographic criteria for success and failure.
Bleeding time | During hemostasis (0-10 minutes)
  Recording the bleeding time of different participants during hemostasis.

SECONDARY OUTCOMES:
Post-operative pain | 24 hours, 3 days, 1 week
  Recording the post-operative pain using Heft-Parker visual analogue scale Minimum value: None Maximum value: Maximum possible The higher values indicate more post-operative pain

CONTACTS AND LOCATIONS:
Locations (1):
- Misr International University, Cairo, Obour, Egypt

IPD SHARING:
Plan to Share IPD: No